CLINICAL TRIAL: NCT00468533
Title: The Monitor of Serum Prolactin Level and Related Clinical Observations Among Individuals With Schizophrenia Spectrum Illnesses in a 3 Months Aripiprazole Trial
Brief Title: The Monitor of Serum Prolactin Level in a 3 Months Aripiprazole Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yu-Li Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YLH-IRB-9506
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2007-05-02 (Estimated); Status verified 2007-04

CONDITIONS: Schizophrenia, Tardive Dyskinesia, Metabolic Syndrome
Keywords: Arupiprazole, prolacin, PANSS, CGI, AIMS
MeSH Terms: conditions — Schizophrenia; Tardive Dyskinesia; Metabolic Syndrome | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
A short term post-market monitoring of serum prolactin level change among patients with schizophrenia shifting from other antispychotics to different dosages of aripiprazole.

DETAILED DESCRIPTION:
This is an open-label clinical trial of adult inpatients or outpatients with a diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder as measured by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR). Eligible patients will have laboratory and clinical assessments completed. All procedures in this study are considered standard care and impose no additional risks to the patients. Participation is voluntary and recruitment will be on an "as come" basis.

Study Visits Schedule

Visit 1 Visit 2 Visit 3 Visit 4 Visit 5 Visit 6 Day -7 Day 7 Day 14 Day 21 Day 28 Day 90 Baseline Initiation Endpoint prolonged f/u

Discussion of Design and Control

Because of the ethical concerns regarding withholding medication from seriously ill patients, this study does not employ a washout period. Though patients may have their antipsychotic drug held for up to 12 hours, this should not present any clinical problems in the majority of patients. This one day prevalence trial allows for clinical data to be collected in a timely manner.

Study Population

Most subjects recruited in this study are originated from a chronic psychiatric residential community. They are characterized by a regular medication with reliable drug compliance under a well-controlled diet in the unit. The subject of drug naïve will be denoted and analyzed separately in the later stage.

Entry Procedures

The patient and/or the patient's authorized legal representative prior to the patient's participation in the study will sign an informed consent document approved by an ethical review board, or similar body.

Inclusion Criteria

Patients may be included in the study if they meet the following criteria:

1. Males and females 16-65 years of age
2. Diagnosis of schizophrenia, schizoaffective or schizophreniform disorder
3. Each individual must have a level of understanding sufficient to perform all tests and examinations required
4. Individuals must be willing to fast after midnight the evening prior to study visit
5. Individuals must be willing to provide a small sample of blood for evaluation
6. Individuals must be willing to participate in a short 30-45 minute clinical interview

Exclusion criteria

Patients may be excluded from the study for any of the following reasons:

1. A current diagnosis of diabetes mellitus
2. Serious unstable illness such that death is anticipated within 1 year or intensive care unit hospitalization for the condition is anticipated within 6 months
3. Uncorrected hypothyroidism or hyperthyroidism
4. Uncorrected tumor secreting ectopic prolactinemia

Dosage and Administration The dosage of aripiprazole will be co-administrated since day 1 with the fixed dosage of 10 mg aripiprazole per day for 1 week with the full dosage of previously used antipsychotics. The previous antipsychotics will be removed on day 8, and each individual will be assigned to either 10-15 mg aripiprazole per day (A arm) or 20-30 mg aripiprazole per day (B arm) or 10mg aripriprazole plus 1mg haldol per day (C arm) via the randomized procedure.

Visit 1 Visit 2 Visit 3 Visit 4 Visit 5 Visit 6 Visit 7 Day -7 Day 7 Day 14 Day 21 Day 28 Day 60 Day 90 Previous antispychotics Full dosage stop - - - A arm (N=16) 10mg 10-15mg 10-15mg 10-15mg 10-15mg 10-15mg B arm (N=16) 10mg 20-30 mg 20-30 mg 20-30 mg 20-30 mg 20-30 mg C arm (N=16) 10mg 10mg (+ 1-2 mg haldol) 10mg (+ 1-2 mg haldol) 10mg (+ 1-2 mg haldol) 10mg (+ 1-2 mg haldol) 10mg (+ 1-2 mg haldol) Denotation: C arm is designed for the purpose of evaluation on add-on effect from typical antipsychotics with a high potency such as haldol. The difference between C arm and the other two might be minimal or significant due to different reaction in Asian population or Chinese population.

In addition to the necessary prescription of antipsychotics described as above listed, adequate amount of benzodiazepines and anticholinergics are permitted to give to alleviate the possible anxiety, insomnia, and EPS as an adjunctive agent simultaneously.

Table 1

Visit 1 Visit 2 Visit 3 Visit 4 Visit 5 Visit 6 Visit 7 Day -7 Day 7 Day 14 Day 21 Day 28 Day 60 Day 90 CGI x x x x x x x DRA x x x x PANSS x x x x AIMS x x x x SAS x x x x SWN x x x x Demographic Sheet x

Clinical Laboratory Tests Clinical laboratory testing will be performed at Visit 1, 2, 3, 4, 5, 6. See Table2 for a complete list of tests to be performed. Patients will be asked to fast after midnight (at least 8 hours) prior to labwork. If a patient is to take morning medications, he/she is asked to hold the morning medications until after the labwork is drawn. He or she may take the medication immediately after the labs have been drawn. Note: A patient is permitted to go off site to have his/her labs drawn. Labwork must be drawn within 3 days of time the demographic and other data is/was gathered.

Table 2

Visit 1 Visit 2 Visit 3 Visit 4 Visit 5 Visit 6 Visit 7 Day -7 Day 7 Day 14 Day 21 Day 28 Day 60 Day 90 Prolactin x x x x x x x Leptin x x x x Estrogen x x x x Glusoce x x x x x x x Insulin x x x x x x x Total cholesterol x x x x HDL x x x x LDL x x x x Triglycerides x x x x

Other Clinical Assessments Hypertension is defined as systolic blood pressure (SBP) of 140 mm Hg or greater, diastolic blood pressure (DBP) of 90 mm Hg or greater, or taking antihypertension medication. Obesity is defined as a Body Mass Index (BMI) of 30 or greater.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study if they meet the following criteria:

1. Males and females 16-65 years of age
2. Diagnosis of schizophrenia, schizoaffective or schizophreniform disorder
3. Each individual must have a level of understanding sufficient to perform all tests and examinations required
4. Individuals must be willing to fast after midnight the evening prior to study visit
5. Individuals must be willing to provide a small sample of blood for evaluation
6. Individuals must be willing to participate in a short 30-45 minute clinical interview

Exclusion Criteria:

Patients may be excluded from the study for any of the following reasons:

1. A current diagnosis of diabetes mellitus
2. Serious unstable illness such that death is anticipated within 1 year or intensive care unit hospitalization for the condition is anticipated within 6 months
3. Uncorrected hypothyroidism or hyperthyroidism
4. Uncorrected tumor secreting ectopic prolactinemia

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-05; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
prolactin level drops after shifting to aripiprazole | 3 months

SECONDARY OUTCOMES:
correlations between prolactin and other clinical outcomes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tsuo-Hung Lan, MD, PhD, Principal Investigator — Yu-Li Hospital
Locations (1):
- Yu-Li Hospital, DOH, Hualien City, Hualien, Taiwan